CLINICAL TRIAL: NCT04897958
Title: Prediction of the PRONOUNCE Prostate Cancer Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-PRONOUNCE
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Degarelix: Reference group
  Interventions: Drug: Degarelix
- Leuprolide: Exposure group
  Interventions: Drug: Leuprolide

INTERVENTIONS:
Drug: Degarelix — Degarelix dispensing claim is used as the reference group.
  Groups: Degarelix
Drug: Leuprolide — Leuprolide dispensing claim is used as the exposure group.
  Groups: Leuprolide

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates:

The degarelix indication for treatment of prostate cancer was approved by the FDA on Dec 24, 2008. Leuprolide was initially approved for the same indication prior to Dec 24, 2008.

IBM MarketScan: Dec 24, 2008 - December 31, 2018 (end of available data) Optum CDM: Dec 24, 2008 - June 30, 2020 (end of available data) CMS Diabetes: Dec 24, 2008 - Dec 31, 2017 (end of available data)

Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Pre-existing ASCVD (confirmed diagnosis, documented) according to a least 1 of the following criteria:
* Previous MI >= 30 days before randomization
* Previous revascularization procedure >= 30 days before randomization
* Coronary artery: stent placement/balloon angioplasty or coronary artery bypass graft surgery
* Carotid artery: stent placement/balloon angioplasty or endarterectomy surgery
* Iliac, femoral, popliteal arteries: stent placement/balloon angioplasty or vascular bypass surgery

Exclusion Criteria:

* Treatment naivety (ADT)
* Previous or current hormonal management of prostate cancer including surgical castration, any hormonal manipulation, or any previous neoadjuvant/adjuvant hormonal therapy, unless treatment was terminated more than 12 months prior to enrollment
* Uncontrolled Type 1 or Type 2 diabetes mellitus
* Uncontrolled hypertension
* A history of congenital long QT syndrome or risk factors for Torsade de pointes ventricular arrhythmias
* MI; stroke; or coronary, carotid, or peripheral artery revascularization

Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Subjects were selected on the basis of having at least one diagnosis code indicating prostate cancer, male sex, and a history of artherosclerotic cardiovascular disease. In contrast to the the PRONOUNCE RCT trial, patients cannot be required to have had established tumor staging information, angiography-verified stenosis/occlusion of vessels, and a lack of planned cardiac surgery at the time of treatment initiation due to poor capture of this information administrative data. All patients were required to have continuous enrollment for 365 days prior to cohort entry to ensure incident use of the study drugs.
Sampling Method: Non-Probability Sample
Enrollment: 14417 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | Through study completion (earliest of 336 days or censoring)
  Composite of all-cause mortality, nonfatal MI, and nonfatal stroke

SECONDARY OUTCOMES:
All-Cause Mortality | Through study completion (earliest of 336 days or censoring)
  Component of MACE
Nonfatal MI | Through study completion (earliest of 336 days or censoring)
  Component of MACE
Nonfatal Stroke | Through study completion (earliest of 336 days or censoring)
  Component of MACE

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT04897958/Prot_SAP_001.pdf